CLINICAL TRIAL: NCT01042665
Title: Relationship Between Intraocular Pressure Fluctuation and Retinal Ganglion Cell Function in Eyes Receiving Latanoprost 0.005% Versus Placebo
Brief Title: Relationship Between Eye Pressure and Ganglion Cell Function in Eyes Receiving Latanoprost Versus Placebo
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, David S. Greenfield, Professor of Ophthalmology, University of Miami
Other Study IDs: 20057259
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Glaucoma
Keywords: Glaucoma; intraocular pressure; latanoprost; retinal ganglion cell; pattern electroretinogram
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- primary open angle glaucoma: Patients with glaucomatous optic neuropathy defined as narrowing of the neuroretinal rim, notching, excavation, or RNFL defect; and repeatable standard automated perimetry abnormality defined as a glaucoma hemifield test (GHT) "outside normal limits" or pattern standard deviation (PSD) outside 95% normal limits were included.
  Interventions: Drug: latanoprost 0.005%; Drug: Placebo
- Ocular Hypertensive group: Ocular hypertension defined as an intraocular pressure ≥ 24 mm Hg and ≤ 32 mm Hg in one eye and IOP ≥ 22 mm Hg and ≤ 32 mm Hg in the fellow eye, with normal optic disc, normal visual field defined as follows mean Deviation (MD) or Pattern Standard Deviation (PSD) of p>5%, normal Glaucoma Hemifield Test (GHT) and reliable visual field exam
  Interventions: Drug: latanoprost 0.005%; Drug: Placebo

INTERVENTIONS:
Drug: latanoprost 0.005% — Active comparator
  Other Names: Xalatan
Drug: Placebo — Placebo comparator
  Other Names: Inactive tear drops

SUMMARY:
The purpose of this investigation is to evaluate the relationship between IOP fluctuation, RGC dysfunction, and optic nerve and retinal nerve fiber layer (RNFL) thickness changes in patients with glaucoma and ocular hypertension receiving latanoprost 0.005% versus placebo.

DETAILED DESCRIPTION:
It has been hypothesized that intraocular (IOP) variability is an independent risk factor for the progression of glaucoma. IOP variability includes 24 hour IOP fluctuation during the waking period (diurnal fluctuation) and sleep period (nocturnal fluctuation) as well as longitudinal IOP variability measured in the diurnal period over the course of multiple office visits.

Latanoprost has been clinically used to lower eye pressure in glaucoma and ocular hypertension for almost 10 years. Latanoprost 0.005% has been demonstrated to provide superior ocular hypotensive efficacy compared with timolol 0.5% in pivotal phase 3 clinical trials (Alm et al. 1995; Camras 1996).

The Pattern Electroretinogram (PERG) is a non-invasive technology that objectively measures the retinal ganglion cell (RGC) function (Porciatti and Ventura 2004). A recent study has demonstrated that the RGC function can be improved following IOP reduction in glaucomatous eyes with early visual field defects (Ventura and Porciatti 2005).

The purpose of this investigation is to evaluate the relationship between IOP fluctuation, RGC dysfunction, and optic nerve and retinal nerve fiber layer (RNFL) thickness changes in patients with glaucoma and ocular hypertension receiving latanoprost 0.005% versus placebo.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - OHT:

* Ocular hypertension defined as an IOP ≥ 24 mm Hg and ≤ 32 mm Hg in one eye and IOP ≥ 22 mm Hg and ≤ 32 mm Hg in the fellow eye
* Normal optic disc
* Normal visual field defined as follows:
* Mean Deviation (MD) or Pattern Standard Deviation (PSD) of p>5%
* Normal Glaucoma Hemifield Test (GHT)
* Reliable visual field exam (less than 33% false positives or false negatives, and less than 20% fixation losses)

Inclusion Criteria - POAG:

* Glaucomatous visual field loss defined as a CPSD (p < 0.05), or GHT (p < 1%) outside normal limits with consistent with ONH or NFL defect
* Early visual field loss defined as MD ≤ -6.0 dB
* Untreated IOP ≤ 32 mmHg
* ONH or NFL defect defined as either inter-eye CDR asymmetry > 0.2, rim thinning or notching, or NFL bundle defect visible on slitlamp biomicroscopy and stereo color fundus photography

Exclusion Criteria:

Exclusion Criteria - OHT:

* Best-corrected visual acuity less than 20/40 either eye
* Abnormal or unreliable VF
* Untreated IOP > 32 mmHg
* Age < 18 or >85 years
* Refractive error of > +3.00 D or < -7.00 D
* Previous intraocular surgery except for uncomplicated cataract extraction with posterior chamber intraocular lens implantation
* Need for chronic ocular or systemic corticosteroid use
* Narrow/closed angle (gonioscopy must show 75% or more of the angle to be Grade 2 or more by Shaffer's grading system)
* Diabetic retinopathy
* Other diseases that may cause VF loss or optic disc abnormalities
* Life-threatening or debilitating illness making it unlikely patient could successfully complete the study
* Inability to clinically view or photograph the optic discs due to media opacity or poorly dilating pupil
* Refusal of informed consent or of commitment to the full length of the study
* Contraindication to latanoprost or placebo vehicle

Exclusion criteria - POAG:

* Best-corrected visual acuity less than 20/40
* Untreated IOP > 32 mmHg
* Age < 18 or >85 years
* Refractive error of > +3.00 D or < -7.00 D
* Previous intraocular surgery except for uncomplicated cataract extraction with posterior chamber intraocular lens implantation
* Diabetic retinopathy
* Other diseases that may cause VF loss or optic disc abnormalities
* Inability to clinically view or photograph the optic discs due to media opacity or poorly dilating pupil
* Inability to perform reliably on automated VF testing
* Life-threatening or debilitating illness making it unlikely patient could successfully complete the study.
* Refusal of informed consent or of commitment to the full length of the study
* Contraindication to latanoprost or placebo vehicle

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary open angle glaucoma or ocular hypertension from the Glaucoma Clinic at Bascom Palmer Eye Institute- Palm Beach Office.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evidence of impact of intraocular (IOP) reduction on retinal ganglion cell (RGC) function | 8 weeks
  RGC function is evaluated by pattern electroretinogram optimized for glaucoma (PERGLA)

CONTACTS AND LOCATIONS:
Overall Officials: David S Greenfield, MD, Principal Investigator — University of Miami Bascom Palmer Eye Institute
Locations (1):
- University of Miami Bascom Palmer Eye Institute, Palm Beach Gardens, Florida, United States